CLINICAL TRIAL: NCT02696447
Title: Radiation Therapy and Venous Thromboembolic Events
Brief Title: Radiation Impact on Thromboembolic Events
Acronym: RIT
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); CH Roanne (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2015-09
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Malignant Neoplasm
Keywords: Radiation therapy; Thrombosis
MeSH Terms: conditions — Neoplasms; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer treated by radiotherapy: Patient with a solid cancer (all locations) treated with radiation therapy and/or brachytherapy as curative intent
  Interventions: Biological: Biomarkers assays

INTERVENTIONS:
Biological: Biomarkers assays — D-Dimer assays, C-reactive protein, blood platelets assays

SUMMARY:
The aim of the present study is to determine the frequency and to identify main risk factors for venous thromboembolism of venous thromboembolic complications in a population of cancer patients treated with a curative intent by ionizing radiation.

ELIGIBILITY:
Inclusion Criteria:

* patient with a solid cancer (all locations) treated with radiation therapy and / or brachytherapy as curative intent
* to be 18

Exclusion Criteria:

* Patient with metastatic cancer,
* Patients whose follow-up at 6 months is not possible
* Patient receiving an anti-coagulative medication (curative doses)
* Pregnant or breastfeeding women,
* Person under protection of justice or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with a solid (all locations) treated with radiation therapy and / or brachytherapy as curative intent
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Venous Thromboembolism event | 6 months
  All venous thromboembolism, whether symptomatic or discovered incidentally, objectified (CT angiography, lung scintigraphy, venous Doppler) between J1 of radiation treatment, up to 6 months following discontinuation of radiation treatment

SECONDARY OUTCOMES:
Dosage of D-dimer | 6 months
C-reactive protein | 6 months
Complete blood count | 6 months
Time of occurrence of VTE | 6 months
  Time of occurrence of VTE
Symptomatic VTE | 6 months
  Symptomatic VTE.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH de Roanne, Roanne
  - Institut de cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daguenet E, Maison M, Tinquaut F, Giroux EA, Bertoletti L, Suchaud JP, Rancoule C, Guy JB, Magne N. Venous thromboembolism and radiation therapy: The final radiation-induced thrombosis study analysis. Cancer Med. 2022 Apr;11(8):1753-1762. doi: 10.1002/cam4.4559. Epub 2022 Feb 24. PMID 35199492